CLINICAL TRIAL: NCT01961895
Title: Evaluation of the Effect of Perioperative Continuous Lumbar Plexus Block Upon the Incidence of Ischemic Cardiovascular Events in Elderly Patients With Hip Fracture.
Brief Title: Lumbar Plexus Block Upon the Incidence of Ischemic Cardiovascular Events in Elderly Patients With Hip Fracture
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pontificia Universidad Catolica de Chile (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Altermatt 09-148
Record Dates: First submitted 2013-10-10; First posted 2013-10-14 (Estimated); Last update posted 2013-10-14 (Estimated); Status verified 2013-10

CONDITIONS: Hip Fractures; Perioperative Myocardial Ischemia
Keywords: Continuous lumbar plexus (LP) block analgesia
MeSH Terms: conditions — Hip Fractures | interventions — Analgesia, Patient-Controlled

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intravenous patient-controlled analgesia (Active Comparator): Intravenous morphine solution 0.2 mg / ml in PCA mode without basal infusion, 1mg bolus demand and lockout of 8 minutes.
  Interventions: Drug: Intravenous patient-controlled analgesia
- Continuous lumbar plexus (LP) block analgesia (Experimental): Continuous lumbar plexus (LP) block analgesia. Continuous infusion of a solution of 0.1% bupivacaine in PCA mode, programmed at 8 ml / h.
  Rescue bolus 5 ml and 30 minutes lockout
  Interventions: Procedure: Continuous lumbar plexus (LP) block analgesia

INTERVENTIONS:
Procedure: Continuous lumbar plexus (LP) block analgesia
  Arms: Continuous lumbar plexus (LP) block analgesia
Drug: Intravenous patient-controlled analgesia
  Arms: Intravenous patient-controlled analgesia

SUMMARY:
The purpose of this study is evaluate the efficacy of perioperative continuous lumbar plexus block in reducing the risk of cardiac ischemic events of elderly patients undergoing surgery for hip fractures, expressed as a reduction of ischemic events per subject.

ELIGIBILITY:
Inclusion Criteria:

* Patients with hip fracture within 48 hours of evolution
* Known coronary artery disease:

Previous myocardial infarction Chronic stable angina Atypical angina with positive exercise test for coronary flow failure. Evidence of coronary artery disease with ultrasound, scintigraphic or angiographic compatible

* Patients with at least two of the risk factors for coronary heart disease as defined by Wallace (1998)

Exclusion Criteria:

* Patients receiving orthopedic treatment.
* Patients with coagulopathy, clinic or laboratory.
* Patients with sepsis or infection of the catheter insertion site of lumbar plexus.
* Patients with neurological diseases evolving.
* Patients disoriented, or dementia.
* CKD stage IV National Kidney Foundation (2)
* Glomerular filtration rate between 15 and 29 mL/min/1, 73 m2
* Patients unable to use the Numeric Rating Scale (NRS) to assess pain.
* Patients with non-sinus rhythm or conduction abnormalities (right bundle branch block or left, atrioventricular block) in the admission ECG
* Patients with pacemaker.
* Enrolled patients with acute coronary syndrome or decompensated cardiovascular disease at entry.
* Allergy to any of the drugs of the protocol.
* Inability to understand or unaided sign informed consent.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2010-05; Primary Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
evaluate the efficacy of perioperative continuous lumbar plexus block in reducing the risk of cardiac ischemic events of elderly patients undergoing surgery for hip fractures, expressed as a reduction of ischemic events per subject. | 3 days

SECONDARY OUTCOMES:
Major cardiovascular events (myocardial infarction, acute pulmonary edema, arrhythmias). | 3 days
hospital death | 3 days
Death at 30, 90 and 360 days after surgery | 1 year
Perioperative Pain Intensity, measured in numerical rating scale (NRS). | 3 days
Evaluate Adverse events (hypotension, respiratory depression, systemic toxicity, etc..) | 3 days

CONTACTS AND LOCATIONS:
Locations (2):
- Chile (2):
  - Division de Anestesia - Pontificia Universidad Catolica de Chile, Santiago, Santiago Metropolitan
  - División de Anestesia - Facultad de Medicina Pontificia Universidad Católica, Santiago, Santiago Metropolitan

REFERENCES:
- [Derived] Guay J, Kopp S. Peripheral nerve blocks for hip fractures in adults. Cochrane Database Syst Rev. 2020 Nov 25;11(11):CD001159. doi: 10.1002/14651858.CD001159.pub3. PMID 33238043